CLINICAL TRIAL: NCT02290899
Title: Modulation of Behavioral Inhibition in Attention Deficit Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: Rhode Island Hospital (Other)
Collaborators: Nancy Lurie Marks Family Foundation (Other); Bradley Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 4067-14
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-04

CONDITIONS: ADHD
Keywords: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

SUMMARY:
The main purpose of this study is to investigate how the brain responds to a procedure known as transcranial direct current stimulation (tDCS) and how tDCS affects performance on a behavioral task. Research suggest that this procedure leads to improvement in brain and behavioral measures of inhibitory control (controlling impulses) in healthy control participants. The investigators want to explore whether the same improvement will be seen in kids with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ADHD
* Parent informed consent and child assent

Exclusion Criteria:

* Intracranial pathology from a known genetic disorder (e.g., Neurofibromatosis Type 1 (NF1), tuberous sclerosis) or from acquired neurologic disease (e.g. stroke, tumor), cerebral palsy, history of severe head injury, or significant dysmorphology
* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, or immediate (1st degree relative) family history epilepsy
* Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
* History of head injury resulting in prolonged loss of consciousness
* Substance abuse or dependence within the past six months
* Chronic treatment with prescription medications that decrease cortical seizure threshold that the patient is unable to withhold from taking during study visits
* Damaged skin on the scalp (i.e., skin with ingrown hairs, acne, razor nicks, wounds that have not healed, recent scar tissue, broken skin, etc.)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with ADHD
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
Stop-Signal Task | Immediately following tDCS

CONTACTS AND LOCATIONS:
Locations (1):
- Bradley Hospital, East Providence, Rhode Island, United States